CLINICAL TRIAL: NCT02544893
Title: Postoperative Analgesic Effects of Using Bupivacaine Alone or Added Dexmedetomidine for Ultrasound Guided Thoracic Paravertebral Block in Thoracotomy
Brief Title: Postoperative Analgesic Effects of Using Dexmedetomidine for Ultrasound Guided Thoracic Paravertebral Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Esra Nur Ünalan, resident, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014/649
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- bupivacaine (Active Comparator): 0,5% 20 ml bupivacaine added 0.9% 1 ml serum physiologic on paravertebral block
  Interventions: Drug: bupivacaine
- dexmedetomidine (Active Comparator): 100 mcg dexmedetomidine added to 0,5% 20 ml bupivacaine on paravertebral block
  Interventions: Drug: dexmedetomidin
- serum phsyologic (Active Comparator): 0,9% 21 ml serum physiologic
  Interventions: Drug: serum physiologic

INTERVENTIONS:
Drug: bupivacaine — 21 ml 0.5 %bupivacaine is applied paravertebral space
  Other Names: marcaine
  Arms: bupivacaine
Drug: dexmedetomidin — 1 ml dexmedetomidin + 20 ml 0.5 % bupivacaine are applied paravertebral space
  Other Names: precedex
  Arms: dexmedetomidine
Drug: serum physiologic — 21 ml serum physiologic is applied paravertebral space
  Arms: serum phsyologic

SUMMARY:
we aimed postoperative analgesic effects of using bupivacaine alone or added dexmedetomidine for ultrasound guided thoracic paravertebral block in thoracotomy

DETAILED DESCRIPTION:
paravertebral block is commonly used in the treatment for acute and chronic pain.The duration of paravertebral block could theoretically be prolonged with neurolytic agents. Dexmedetomidine ,an alfa-2 adrenoreceptor agonist, is being used and adjuvant capable of prolonging duration of sensory and motor block on nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* 18-65 aged
* patient undergoing thoracotomy

Exclusion Criteria:

* chronic opioid consumption
* bupivacaine and dexmedetomidine allergies
* coagulopathy
* infection at the needle insertion side
* chronic liver and kidney disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
opioid consumption | postoperative 24 hours
  patient controlled analgesia

SECONDARY OUTCOMES:
visual analog scale | postoperative 1 day
  visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: esra n ünalan, resident, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University Medicine Faculty, Kayseri, Turkey (Türkiye)